CLINICAL TRIAL: NCT02273544
Title: Bioavailability of Dipyridamole After Asasantin (Extended Release 200mg Dipyridamole/25mg ASA) in 3 Experimental Formulations (Given b.i.d. Over 3 or 5 Days, Respectively) Relative to the Standard Formulation in 16 Healthy Female and Male Subjects. Intraindividual Comparison, Randomised, Open
Brief Title: Study to Evaluate Pharmacokinetics of Dipyridamole in Three New Formulations of Asasantin ER in Healthy Female and Male Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 9.158
Record Dates: First submitted 2014-10-23; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (4):
- Asasantin ER (new formulation - low) (Experimental)
  Interventions: Drug: Asasantin ER (new formulation - low)
- Asasantin ER (new formulation - medium) (Experimental)
  Interventions: Drug: Asasantin ER (new formulation - medium)
- Asasantin ER (new formulation- high) (Experimental)
  Interventions: Drug: Asasantin ER (new formulation - high)
- Asasantin ER - commercial formulation (Active Comparator)
  Interventions: Drug: Asasantin ER - commercial formulation

INTERVENTIONS:
Drug: Asasantin ER (new formulation - low)
  Arms: Asasantin ER (new formulation - low)
Drug: Asasantin ER (new formulation - medium)
  Arms: Asasantin ER (new formulation - medium)
Drug: Asasantin ER (new formulation - high)
  Arms: Asasantin ER (new formulation- high)
Drug: Asasantin ER - commercial formulation
  Arms: Asasantin ER - commercial formulation

SUMMARY:
The objective of this study was to compare the pharmacokinetics of dipyridamole in three different Asasantin ER batches (test) containing different amounts of retarding lacquers to the existing commercial product at steady state with b.i.d. treatment

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects as determined by results of screening
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Female subjects are not lactating. Females must use adequate contraception (adequate contraception e.g. sterilization, IUP, oral contraceptives) prior to administration of study medication, during the study until after release from the study. Women must have negative blood pregnancy tests
* Age >= 18 and <= 60 years
* BMI >=18.5 and <=29.9 kg/m2 (see abbreviations for formula)
* Able to communicate well with the investigator and to comply with study requirements
* Laboratory values within a clinically defined reference range

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate, and electrocardiogram) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which were deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) (< 1 month prior to administration or during the trial)
* Use of any drugs, which might influence the results of the trial, (< 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (< 1 months prior to administration (at least 10 times the relevant elimination half-life) or during trial)
* Having had prescription medication 2 weeks prior to study drug administration or over the counter medication 1 week prior to study drug administration (at least 10 times the relevant elimination half-life)
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day)
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Use of methylxanthine-containing drinks or foods (coffee, tea, cola, energy drinks, chocolate, etc.), grapefruit or grapefruit juice, alcohol, green tea, or tobacco < 5 days prior to administration of study drug
* Blood donation or loss > 400 mL (< 1 month prior to administration or during the trial)
* Excessive physical activities (< 5 days prior to administration or during the trial)
* Any ECG value outside of the reference range of clinical relevance including, but not limited to QTcB > 480 ms or QRS interval > 110 ms
* History of any familial bleeding disorder
* Inability to comply with dietary regimen of study centre
* Inability to comply with investigator's instructions

For Female Subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception (adequate contraception e.g. sterilization, Intrauterine Pessary (IUP), oral contraceptives)
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

During the interval between screening and start of drug administration tobacco and caffeine are restricted to avoid withdrawal when starting medication. As no relevant influence on Pharmacokinetic parameters is known moderate tobacco and caffeine consumption are allowed to facilitate trial participation (up to 10 cigarettes or 3 cigars or 3 pipes/day, and/or up to three cups of coffee respectively). Ovarian hormone substitution and oral contraception are allowed to be continued during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2002-09; Primary Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Urinary excretion of dipyridamole | day 2, day 3
  geometric means of percentage of amount excreted from time zero to 10 h (% Ae 0-10h)

SECONDARY OUTCOMES:
Cmax urine (Maximum measured concentration of the analyte) | 0 to 3 hours after drug intake
  Urine collected fraction from 0 -3 hours as surrogate for Cmax
Cmin (Minimum measured concentration of the analyte) | 8 - 10 hours after drug intake
  Urine collected fraction from 8 - 10 hours as surrogate for Cmin
% PTF urine (peak trough fluctuation) | Up to 10 hours after drug intake
  Estimated from the difference of percentage amount excreted from 1 - 3 hours (%Ae (1-3hours) and %Ae (8-10 hours) divided by the average excretion rate over the total dosing interval
Number of subjects with adverse events | up to 1 month